CLINICAL TRIAL: NCT05222230
Title: FFP3 Respirators and Ears - Effects on Middle Ear Pressure and Hearing
Acronym: FFP3-RAE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SP0620
Record Dates: First submitted 2021-09-20; First posted 2022-02-03 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2021-10

CONDITIONS: Eustachian Tube Dysfunction; Hearing Disorders; Nasal Obstruction
Keywords: FFP3M respirators; eustachian tube dysfunction; hearing loss; audiometry; tympanometry
MeSH Terms: conditions — Hearing Disorders; Nasal Obstruction; Hearing Loss

STUDY DESIGN:
Intervention Model Description: Prospective open label basic science study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FFP3 Respirator (Experimental): Participants will wear FFP3 respirators during the study.
  Interventions: Other: FFP3 Mask

INTERVENTIONS:
Other: FFP3 Mask — Participans will wear FFP3 respirators during the study.

SUMMARY:
This is Prospective Basic Science Study whose aims are as follows:

1. To determine the effect of Filtering Facepiece (FFP3M) respirators on eustachian tube function and hearing
2. To evaluate the extent to which FFP3M respirators attenuate speech in decibels

The outcome measures are as follows:

1. Changes in baseline pure tone audiometry and tympanometry post intervention.
2. SNOT-22 Questionnaires before and after use of respirator
3. ETDQ7 questionnaire
4. Measurement of speech attenuation in decibels.

DETAILED DESCRIPTION:
The use of facemasks is one of the key strategies for reducing human to human transmission of SARS-CoV-2. There is a variety of facemasks worn in the clinical environment ranging from simple facemasks to devices such as filtering face piece 3M (FFP3M) respirators which are mandatory for some clinicians performing aerosol generating procedures (AGPs.)

It has been shown that wearing face protective equipment attenuates sound causing decay in speech intelligibility, especially transmission of middle-to-high voice frequencies.It has been shown that wearing surgical masks results in up to 23.3% loss of speech intelligibility in noisy environments with advanced face personal protective equipment such as FFP3M devices, accounting for up to 69.0% reduction of speech intelligibility. A reduction in speech intelligibility leads to reduced understanding which may result in miscommunication thereby compromising patient safety. To date, there have been two critical incidents in our department due to miscommunication attributed to wearing FFP3M respirators.

Anecdotally, clinicians have reported nasal congestion and subjective hearing loss during FFP3M respirator usage and after, especially when they are worn for a prolonged period of time. Clinicians working in theatre may be required to wear these devices for a number of hours when involved with AGPs.

The secondary consequences of wearing FFP3M respirators for prolonged periods of time, especially in a theatre setting require scientific exploration. This study aims to investigate the effect of FFP3M respirators on middle ear pressure and hearing, and the extent to which FFP3M respirators attenuate sound. Investigators believe that a reduction in speech intelligibility is not the only explanation for the perception of hearing loss when using FFP3M respirators. Investigators postulate that a transient dysfunction in the eustachian tube pressure regulating system also contributes to hearing loss.

To test this hypothesis, investigators will measure hearing and middle ear pressure using pure tone audiometry and tympanometry before and during FFP3M usage. Investigators will also use SNOT-22 and ETDQ7 questionnaires which are validated patient reported outcome measures for nasal symptoms and eustachian tube function. Investigators hope that this study provides some understanding of the physiological effects of FFP3M respirators on hearing and sinonasal symptoms and improves our understanding of their impact on clinical practice. There are no current studies looking into the effects of FFP3M respirators on eustachian tube function.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers that already have their own masks, fitted and provided by the Trust for day-to-day clinical use
* Participants without pre-existing sinonasal symptoms or previous sinonasal surgery
* Participants without pre-existing hearing loss or a history of otological procedures

Exclusion Criteria:

* Participants with pre-existing sinonasal symptoms or previous sinonasal surgery
* Participants with pre-existing hearing loss or a history of otological procedures
* Participants who do not satisfy the requirements set out in the pre-registration questionnaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-07-23 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in baseline pure tone audiometry post intervention. | 48 hours
  We will measure changes in baseline pure tone audiometry post FFP3 respirator usage..
Measurement of speech attenuation in decibels. | 1 hours
  We will measure speech attenuation in decibels when participants are wearing FFP3 respirators
Changes in baseline tympanometry post intervention | 48 hours
  We will measure changes in baseline tympanometry post FFP3 respirator usage.

SECONDARY OUTCOMES:
Eustachian tube function | 48 hours
  Participants will complete the SINO-NASAL OUTCOME TEST (SNOT-22) Questionnaire which is a 22 point questionnaire. Participants will be asked to grade the severity of their symptoms from 1-5 with with higher scores denoting severe symptoms.
  The questionnaires will be completed pre and post interventions to investigate changes in eustachian tube function.
Eustachian tube function | 48 hours
  Participants will complete the Eustachian Tube Dysfunction Questionnaire (ETDQ-7) which is a 7 point questionnaire. Patients are asked to grade the severity of their symptoms from 1-7 with with higher scores denoting severe symptoms.
  The questionnaires will be completed pre and post interventions to investigate changes in eustachian tube function.

IPD SHARING:
Plan to Share IPD: No
No data will be shared with other researchers

REFERENCES:
- [Background] Corey RM, Jones U, Singer AC. Acoustic effects of medical, cloth, and transparent face masks on speech signals. J Acoust Soc Am. 2020 Oct;148(4):2371. doi: 10.1121/10.0002279. PMID 33138498
- [Background] Muzzi E, Chermaz C, Castro V, Zaninoni M, Saksida A, Orzan E. Short report on the effects of SARS-CoV-2 face protective equipment on verbal communication. Eur Arch Otorhinolaryngol. 2021 Sep;278(9):3565-3570. doi: 10.1007/s00405-020-06535-1. Epub 2021 Jan 3. PMID 33389012
- [Background] Hampton T, Crunkhorn R, Lowe N, Bhat J, Hogg E, Afifi W, De S, Street I, Sharma R, Krishnan M, Clarke R, Dasgupta S, Ratnayake S, Sharma S. The negative impact of wearing personal protective equipment on communication during coronavirus disease 2019. J Laryngol Otol. 2020 Jul;134(7):577-581. doi: 10.1017/S0022215120001437. Epub 2020 Jul 28. PMID 32641175
- [Background] Hopkins C, Gillett S, Slack R, Lund VJ, Browne JP. Psychometric validity of the 22-item Sinonasal Outcome Test. Clin Otolaryngol. 2009 Oct;34(5):447-54. doi: 10.1111/j.1749-4486.2009.01995.x. PMID 19793277
- [Background] McCoul ED, Anand VK, Christos PJ. Validating the clinical assessment of eustachian tube dysfunction: The Eustachian Tube Dysfunction Questionnaire (ETDQ-7). Laryngoscope. 2012 May;122(5):1137-41. doi: 10.1002/lary.23223. Epub 2012 Feb 28. PMID 22374681